CLINICAL TRIAL: NCT02551224
Title: A Randomized, Open-label, Cross-over Study Comparing the Preference on the Feedback Mechanisms of Dose Delivery Confirmation With the Breezhaler® Device Compared to the Ellipta® Device in Patients With Chronic Obstructive Pulmonary Disease (COPD): The Advantage Study
Brief Title: Preference on the Feedback Mechanisms of Dose Delivery Confirmation With the Breezhaler® Device Compared to the Ellipta® Device in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: Advantage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CQVA149A2405
Record Dates: First submitted 2015-08-31; First posted 2015-09-16 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive (COPD)
Keywords: COPD
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: open-label, cross-over study comparing the preference on the feedback mechanisms of dose delivery confirmation with the Breezhaler® device compared to the Ellipta® device
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breezhaler, then Ellipta (Experimental): Half of the patients will be assigned to first receive a single dose of placebo via the Breezhaler® followed by a single dose of placebo via the Ellipta® inhalation device. The evaluation questionnaires after using each device.
  Interventions: Other: Patient preference questionnaire
- Ellipta, then Breezhaler (Experimental): Half of the patients will be assigned to first receive a single dose of placebo via the Ellipta® followed by a single dose of placebo via the Breezhaler® inhalation device. The evaluation questionnaires after using each device.
  Interventions: Other: Patient preference questionnaire

INTERVENTIONS:
Other: Patient preference questionnaire — The primary variable will be the mean score of questions 1(a) to 1(c) from the preference questionnaire completed at the end of study.

SUMMARY:
The purpose of this study is to compare in COPD patients naïve to DPIs, the perception of the Breezhaler® and Ellipta® devices' feedback mechanisms evaluated using a preference questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of COPD (mild to very severe disease) based on post-bronchodilator FEV1 values in patients with FEV1/FVC <0.70.
* No previous use of DPI.
* Over and either be current smokers or have a history of smoking >10 years. (e.g., 10 pack years = 1 pack/day × 10 years, ½ pack/day × 20 years, etc.):

  * Note: A pack of cigarettes is equal to 20 cigarettes. Occasional smoking of cigars is not relevant to smoking history.
  * An ex-smoker is defined as a patient who has not smoked for ≥6 months at screening.
* Willing and able to reproducibly perform spirometry and inhalational manoeuvers as required by the protocol.
* Willing and able to comprehend and follow the instructions for use of the inhalational devices to be tested in the study.
* Questions or requests for clarification regarding the eligibility of a particular patient based on the above inclusion criteria should be directed to the medical monitor before the patient is enrolled.

Exclusion Criteria:

* History of hypersensitivity to the components of the placebo used in the study or to compounds of similar chemical classes. This includes (but is not exhaustive) patients with known lactose allergy, allergy to magnesium stearate, and those who have suffered paradoxical bronchospasm on inhalation of placebo medications.
* Patients who received treatment with systemic corticosteroids, antibiotics, or had a history suggestive of acute COPD exacerbation and/or hospitalization within 12 weeks prior to the screening or during the baseline period.
* Pregnant or nursing (lactating) women, defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS:

  * Women with reliable contraception methods.
  * Post-menopausal women with no possibility of becoming pregnant.
  * Note: Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to baseline. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Patients with a history (at Visit 1) of asthma indicated by (but not limited to):
* Onset of respiratory symptoms suggestive of asthma (such as cough, wheezing, shortness of breath) prior to age 40.

  • History of a diagnosis of asthma.
* Patients with allergic rhinitis who use an H1 antagonist or intra-nasal corticosteroids intermittently (Treatment with a stable dose or regimen is permitted).
* History of clinically significant conditions including: significant cardiovascular disease, uncontrolled diabetes, a history of non-compliance, alcohol or drug abuse, any patient with active cancer, or any condition in the opinion of the investigator that makes the patient unsuitable for participation in this study.
* Use of investigational drugs (approved or unapproved) in the 3 months before screening.
* Within the 7 days prior to the visits, an increase in episodic use of rescue bronchodilator more than double the average number of puffs used in the preceding week or more than 8 puffs of SABA on any 3 consecutive days or more than 12 puffs of SABA on any 2 consecutive days.
* Respiratory tract infections (sinus, middle ear, oropharyngeal, upper or lower respiratory tract infection) within the 4weeks before the visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Argentina (8):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Vicente López, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Ciudad Autonoma de Bs As

REFERENCES:
- [Derived] Altman P, Bergna MA, Garcia GR, Guerin T, Pino AV, Whiteford JL. Patient perception of Breezhaler(R) and Ellipta(R) device feedback mechanisms in COPD: The ADVANTAGE Study. Curr Med Res Opin. 2019 Feb;35(2):221-227. doi: 10.1080/03007995.2018.1464437. Epub 2018 May 15. PMID 29649916

RESULTS

PARTICIPANT FLOW:
Groups:
- Breezhaler, Then Ellipta group1: Half of the patients will be assigned to first receive a single dose of placebo via the Breezhaler® followed by (minimum of 5 minutes) a single dose of placebo via the Ellipta® inhalation device. The evaluation questionnaires are administered after using each device.
- Ellipta Then, Breezhaler Group 2: Half of the patients will be assigned to first receive a single dose of placebo via the Ellipta® followed by (minimum of 5 minutes) a single dose of placebo via the Breezhaler® inhalation device. The evaluation questionnaires administered after using each device.
Period: First Intervention
Arm/Group | Breezhaler, Then Ellipta group1 | Ellipta Then, Breezhaler Group 2
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Second Intervention (5 Min After First )
Arm/Group | Breezhaler, Then Ellipta group1 | Ellipta Then, Breezhaler Group 2
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 100 subjects were randomized, all of whom were included in the FAS and the safety set
Groups:
- Overall: Half of the patients will be assigned to first receive a single dose of placebo via the Breezhaler® followed by (minimum of 5 minutes) a single dose of placebo via the Ellipta® inhalation device. The evaluation questionnaires were administered after using each device.
Arm/Group | Overall
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 64

OUTCOME MEASURES:

1. Primary Outcome: Patient's Preference on the Feedback Mechanisms of Dose Delivery Confirmation Using the Breezhaler® and Ellipta® Devices
Description: This study will measure patient's perceptions of dose delivery, using a preference questionnaire on use of the Breezhaler® & Ellipta® devices, in COPD patients naïve to DPI devices.The mean (SD) score on a scale of 1- 5 (1 = not at all confident/not at all; 5 = extremely confident/a very great deal) 1a. How confident were you that you received the full dose of medication from your inhaler?
  1=Not At All Confident, 2=Not Very Confident, 3=Somewhat Confident, 4=Confident, 5=Extremely Confident
  1b. How certain were you that there was no drug remaining in the device?
  1=Not At All Certain,2=Not Very Certain, 3=Somewhat Certain,4=Certain, 5=Extremely Certain
  1c. To what extent did the device help you to know that you have received all the medication?
  1=Not At All, 2=A Little, 3=Somewhat, 4=Very Much, 5=A Very Great Deal
Time Frame: 6 hours
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Breezhaler: Half of the patients will be assigned to first receive a single dose of placebo via the Breezhaler® followed by (minimum of 5 minutes) a single dose of placebo via the Ellipta® inhalation device. The evaluation questionnaires were administered after using each device.
- Ellipta: Half of the patients will be assigned to first receive a single dose of placebo via the Ellipta® followed by (minimum of 5 minutes) a single dose of placebo via the Breezhaler® inhalation device. The evaluation questionnaires were administered after using each device.
Arm/Group | Breezhaler | Ellipta
Number analyzed (Participants) | 100 | 100
units on a scale | 4.3 (0.82) | 3.6 (1.05)
Statistical Analysis 1: Comparison: Breezhaler vs Ellipta; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.75, 95% CI 2-sided [0.51 to 0.99]

2. Secondary Outcome: Comfort of the Mouth Pieces for Performing a Tight Seal With the Lips.
Description: To measure in COPD patients naïve to DPIs, the comfort of the mouth pieces when performing a tight seal with the lips using the Breezhaler® and Ellipta® devices.The mean (SD) score on a scale of 1 - 5 (1 = not at all easy, 2= not very easy, 3=somewhat easy, 4=very easy, 5 = extremely easy)
Time Frame: 6 hours
Population: full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breezhaler | Ellipta
Number analyzed (Participants) | 100 | 100
units on a scale | 4.3 (0.70) | 3.9 (0.84)
Statistical Analysis 1: Comparison: Breezhaler vs Ellipta; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.41, 95% CI 2-sided [0.21 to 0.61]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Breezhaler | Ellipta
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 1/100 | 0/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breezhaler (N=100) | Ellipta (N=100)
rhinitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e.,data from all sites)in the clinical trial.